CLINICAL TRIAL: NCT05853874
Title: Sustainable Eating Pattern to Limit Malnutrition in Older Adults
Brief Title: Development of Sustainable Eating Pattern to Limit Malnutrition in Older Adults
Acronym: SENIOR
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: University of Pavia (Other)
Collaborators: Fondazione Salvatore Maugeri (Other); Fondazione IRCCS Policlinico San Matteo di Pavia (Other)
Responsible Party: Principal Investigator, Hellas Cena, Pro-Rector for Third Mission; Professor of Dietetics and Clinical Nutrition; Human Nutrition Researcher and Head of the Clinical Nutrition Laboratory, University of Pavia
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 22042023; CUP: F13C22001210007 (Other Grant/Funding Number: PNRR - MUR)
Record Dates: First submitted 2023-04-26; First posted 2023-05-11 (Actual); Last update posted 2023-05-11 (Actual); Status verified 2023-05

CONDITIONS: Malnutrition; Sarcopenia
Keywords: Nutrition intervention; older adults; malnutrition; sustainability; 24-h recall; sarcopenia; nutritional protocol
MeSH Terms: conditions — Malnutrition; Sarcopenia | interventions — Diet Therapy

STUDY DESIGN:
Intervention Model Description: Randomized Control Trial with two parallel arms. The intervention group will receive a nutritional protocol and the control group will receive the standard of care
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Nutritional intervention (Experimental): Nutritional intervention consist in a macro- and micronutrients balanced nutritional protocol with a focus on sustainability and personalized according to the individual malnutrition severity. In particular, an adequate coverage of energy, protein and water requirements will be guaranteed according to Italian reference values (LARN) and European (ESPEN) guidelines.
  In light of the scientific literature and the principal issues founding in malnourished older people, the proposed nutritional protocol will provide an adequate and sustainable consumption of animal and vegetable proteins and an appropriate water intake.
  The nutritional intervention will be carried out by a qualified staff.
  Interventions: Other: Nutrition intervention (dietary protocol)
- Control (Other): The control group receive the standard of care provided for malnutrition treatment by hospitals
  Interventions: Other: Hospital standard of care

INTERVENTIONS:
Other: Nutrition intervention (dietary protocol) — The nutrition intervention sought to improve participants' overall diet quality, taking into account a sufficient intake of carbohydrates, lipids, fibres and micronutrients (vitamins and minerals), promoting proper fruits and vegetables consumption and variety. About water intake, considering the high dehydration risk in older persons highlighted by the European Society for Clinical Nutrition and Metabolism (ESPEN) guidelines, its adequate consumption is recommended and encouraged.
  Arms: Nutritional intervention
Other: Hospital standard of care — The standard clinical procedures following the malnutrition diagnoses will be implemented according to the routine of the two hospitals
  Arms: Control

SUMMARY:
The SENIOR STUDY is aimed at improving the condition of older adults and malnutrition management in and out Italian hospital settings, since malnutrition is highly prevalent, clinically relevant and potentially treatable conditions. This study consist of two phases: an initial cross-sectional phase and a secondary nutritional intervention phase (RCT).

The SENIOR RCT aim to evaluate the efficacy of a 6 months nutrition protocol intervention compared to hospital standard care on malnourished older adults. Physical and nutritional status will be evaluated through anthropometric measures, blood exams and physical performance. In addition, the individual health perception will be evaluated.

It is expected to find an improvements of the physical and nutritional status.

DETAILED DESCRIPTION:
The SENIOR RCT is a multicenter study conducted in two North Italian Scientific Hospitalization and Treatment Institution in Pavia on older malnourished adults (≥ 65 years old). The estimated duration is 24 months, which include 6 months of nutritional intervention and a follow-up after 6 months, with an preferred starting date on January 2024.

The primary objective of the SENIOR RCT is the evaluation of the efficacy of a 6 months sustainable nutrition protocol on malnourished older adults participants (diagnosed with the most recent GLIM criteria) in comparison to the hospital standard of care.

Therefore, the primary endpoint is the improvement of the nutritional status between pre- and post-intervention between experimental and control group measuring the change of body weight and strength (handgrip).

Secondary objectives are the change pre- and post-intervention between experimental and control group for blood biomarkers, dietary habits, quality of life and evaluation of sarcopenia.

Secondary endpoints are the change pre- and post-intervention between experimental and control group for blood biomarkers, MEDI-LITE score, SF-12, diet composition, phase angle and gait speed.

Participants of this study are older adults over 65 previously enrolled in the SENIOR cross-sectional study and willing to participate to the RCT phase or new enrolled patients from the two hospitals in according to the eligible criteria. Malnutrition will be diagnosed according to GLIM criteria, using Malnutrition Universal Screening Tool (MUST) as screening tool.

The experimental group at the baseline will receive a nutritional assessment followed by the elaboration of a sustainable and personalized nutritional protocol by qualified dietitians. The intervention will last 6 months with a monthly evaluation of the dietary consumption of the previous 24 hour (recall-24h), followed by a final follow-up after additional 6 months.

For both groups at the baseline will be measured blood biomarkers, anthropometric variables, Mediterranean diet adherence, quality of life, strength (handgrip) and locomotion (gait speed). At 3 months weight and strength will be evaluated. At 6- and 12-months baseline measurements will be repeated except for the nutritional assessment.

Dietary habits will be evaluated through a Mediterranean diet questionnaire (MEDI-LITE), while quality of life will be measured with Short-Form Health Survey (SF-12) questionnaire. Anthropometric variables include weight, height (knee height and demi-span), waist circumference, and body composition (BIA). In addition, strength (handgrip) and locomotion (gait speed) will be evaluated. Strength (handgrip), Appendicular Skeletal Mass (ASM) and locomotion (gait speed) are necessary to diagnose sarcopenia according to the European Working Group on Sarcopenia in Older People 2 (EWGSOP2) consensus. Malnutrition will be evaluated again at 6 months.

Blood analysis will be carried out on a subgroup to evaluate the participants' inflammatory, nutritional and clinical status.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 65 years old
* Admission to two Scientific Hospitalization and Treatment Institutions in Pavia, Italy
* Informed consent written and signed
* Malnutrition (GLIM diagnosis)

Exclusion Criteria:

* Dysphagia
* Prior nutritional medical treatment
* Terminal disease
* History of gastric bypass, anorexia nervosa, liver failure
* Dementia or severe confusion (MMSE score<24/30)
* Patients with tumor diagnosis not in remission and currently not treated with oncological therapy
* Patients with chronic or acute respiratory failure
* Barthel index score < 70/100

Ages: 65 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 128 (Estimated)
Dates: Start 2024-01 (Estimated); Primary Completion 2026-01 (Estimated); Study Completion 2026-01 (Estimated)

PRIMARY OUTCOMES:
Change in nutritional status pre- and post- intervention between experimental and control group measuring weight | 24 months (baseline, 3 months, 6 months and 12 months)
  Weight gain= + 2kg
Change in nutritional status pre- and post- intervention between experimental and control group measuring strength | 24 months (baseline, 3 months, 6 months and 12 months)
  Increase in strength = + 1 kg

SECONDARY OUTCOMES:
Changes pre- and post- intervention between experimental and control groups for complete blood count | 24 months (baseline and 6 months)
  Red blood cells (10^9/L), white blood cells (10^12/L or %), hemoglobin (g/dl), hematocrit (%), platelets (10^9/L).
Changes pre- and post- intervention between experimental and control groups for blood lipid profile | 24 months (baseline and 6 months)
  low density lipoprotein (mmol/l), high density lipoprotein (mg/dl), total colesterol (mg/dl), triglicerydes (mg/dl)
Changes pre- and post- intervention between experimental and control groups for blood C reactive Protein (CRP) | 24 months (baseline and 6 months)
  C reactive Protein (CRP) (mg/dl)
Changes pre- and post- intervention between experimental and control groups for blood transaminases | 24 months (baseline and 6 months)
  (glutamic oxaloacetic transaminase, Glutamic-Pyruvic Transaminase, gamma-glutamyl transferase) (U/I) Alkaline phosphatase (U/L)
Changes pre- and post- intervention between experimental and control groups for blood creatin Kinase | 24 months (baseline and 6 months)
  Creatin Kinase (UI/L)
Changes pre- and post- intervention between experimental and control groups for blood prealbumin | 24 months (baseline and 6 months)
  prealbumin (g/mL)
Changes pre- and post- intervention between experimental and control groups for blood cytokine | 24 months (baseline and 6 months)
  interleukin-1β, interleukin-6, interleukin-10, tumor necrosis factor-α, transforming tumor factor-β (pg/ml)
Changes pre- and post- intervention between experimental and control groups for glycemia. | 24 months (baseline and 6 months)
  glycemia (mg/dl)
Changes pre- and post- intervention between experimental and control groups for blood insulin | 24 months (baseline and 6 months)
  Insulin (µU/mL)
Changes pre- and post- intervention between experimental and control groups for blood homocysteine | 24 months (baseline and 6 months)
  Homocysteine (µmol/L)
Changes pre- and post- intervention between experimental and control groups for blood vitamine D | 24 months (baseline and 6 months)
  vitamine D (ng/ml)
Changes pre- and post- intervention between experimental and control groups for blood vitamine B12 | 24 months (baseline and 6 months)
  vitamine 12 (pg/ml)
Changes pre- and post- intervention between experimental and control groups for blood vitamine B9 | 24 months (baseline and 6 months)
  vitamine 9 (ng/mL)
Changes pre- and post- intervention between experimental and control groups for blood sodium (Na) | 24 months (baseline and 6 months)
  Na (mmol/L)
Changes pre- and post- intervention between experimental and control groups for blood potassium (K) | 24 months (baseline and 6 months)
  K (mEq/l)
Changes pre- and post- intervention between experimental and control groups for blood magnesium (Mg) | 24 months (baseline and 6 months)
  Mg (mEq/l)
Changes pre- and post- intervention between experimental and control groups for blood calcium (Ca) | 24 months (baseline and 6 months)
  Ca (mg/dL)
Changes pre- and post- intervention between experimental and control groups for blood iron (Fe) | 24 months (baseline and 6 months)
  Fe (μg)
Changes pre- and post- intervention between experimental and control groups for blood zinc (Zn) | 24 months (baseline and 6 months)
  Zn (mmol/l)
Changes pre- and post- intervention between experimental and control groups for adherence to Mediterranean Diet | 24 months (baseline, 6 months and 12 months)
  Medi-Lite adherence score.score ranges between 0-18. A high score represents a higher adherence to Mediterranean diet.
Changes pre- and post- intervention between experimental and control groups for the quality of life | 24 months (baseline, 6 months and 12 months)
  Short-Form Health Survey 12. Total score ranges between 0-100. A higher score represents a better quality of life
Changes pre- and post- intervention between experimental and control groups for the dietary nutritional composition | 24 months (baseline, 1 month, 2 months, 3 months, 4 months, 5 months, 6 months, 12 months)
  Improvements of dietary composition evaluated with monthly 24-h recalls
Changes pre- and post- intervention between experimental and control groups of fat free mass | 24 months (baseline, 6 months and 12 months)
  Improvement of the phase angle (θ) measured by bioimpedance analysis
Changes pre- and post- intervention between experimental and control groups in locomotion test | 24 months (baseline, 6 months and 12 months)
  Velocity walking increase measured with gait speed test

CONTACTS AND LOCATIONS:
Overall Officials: Hellas Cena, Prof, Principal Investigator — Laboratory of Dietetics and Clinical Nutrition, Department of Public Health, Experimental and Forensic Medicine, University of Pavia; Clinical Nutrition and Dietetics Service, Unit of Internal Medicine and Endocrinology, Pavia; Flavia Magri, Prof, Principal Investigator — Department of Internal Medicine and Therapeutics, University of Pavia and Istituti Clinici Scientifici Maugeri IRCCS, Unit of Internal Medicine and Endocrinology; Istituti Clinici Scientifici Maugeri IRCCS, Unit of Endocrinology and Metabolism, Pavia; Antonio Di Sabatino, Prof, Principal Investigator — Department of Internal Medicine and Therapeutics, University of Pavia; Fondazione IRCCS Policlinico San Matteo, Internal Medicine Unit, Pavia